CLINICAL TRIAL: NCT04512300
Title: Parental Attitude Toward Children Dental Treatment and Care During COVID-19 Pandemic (Cross -Sectional Study)
Brief Title: Parental Attitude Toward Children Dental Treatment During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed Yousry, lecturer in pediatric dentistry Cairo university, Cairo University
Other Study IDs: Covid -19 and dental visit
Record Dates: First submitted 2020-08-12; First posted 2020-08-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Dental Diseases
Keywords: Covid -19; Dental treatment; Dental Care; parental attitude
MeSH Terms: conditions — Stomatognathic Diseases; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is assessment of parental attitude toward children dental treatment and care during Covid 19- crisis

DETAILED DESCRIPTION:
The recent spread of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and its associated coronavirus disease has gripped the entire international community and caused widespread public health concerns.

Many countries all over the world including Egypt, have followed guidelines of limiting dental treatment for emergency cases only. However, as social distancing guidelines are starting to relax across many countries nowadays , dental offices start to reopen for elective procedures , many parents may still have a great concern regarding their children dental treatment during this pandemic. so the aim was to assess their attitude regarding their children dental visit

ELIGIBILITY:
Inclusion Criteria:

* Egyptian parents living in Egypt having children less than 16 years old

Exclusion Criteria:

* incomplete questionnaire

Ages: 1 Year to 16 Years | Sex: All
Age Groups: Child
Study Population: Egyptian parents living in Egypt having children less than 16 years old
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Assessment of parental attitude toward children dental visit during Coronavirus crisis | 10 days
  To assess Egyptian parental attitude toward children dental treatment and care during the current Covid 19- Pandemic. outcome will be measured by questionnaire without scale

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Mohamed, Principal Investigator — Cairo University
Locations (1):
- faculty of dentistry, Cairo university , Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided